CLINICAL TRIAL: NCT07109219
Title: A Modular Phase I/II, Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of AZD4512 Monotherapy or in Combination With Anticancer Agent(s) in Participants With Acute Lymphoblastic Leukemia
Brief Title: Study of AZD4512 Monotherapy or in Combination With Anticancer Agents in Participants With Acute Lymphoblastic Leukemia
Acronym: ALLight
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9891C00001; 2025-522372-93-00 (Other: EU CT number)
Record Dates: First submitted 2025-07-07; First posted 2025-08-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: Acute lymphoblastic leukemia (B-ALL); Dose escalation; Dose optimization; Cluster of differentiation 22 (CD22); Antibody-drug conjugate (ADC)
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1 Dose Escalation (Experimental): Module 1 will evaluate escalating doses of AZD4512 as monotherapy to determine the maximum tolerated dose (MTD) and/or doses of AZD4512 for subsequent evaluation in Module 2 (dose optimization), in participants with relapsed/refractory (R/R) Philadelphia chromosome positive (Ph[+]) and negative (Ph[-]) B-ALL, R/R as defined by National Comprehensive Cancer Network (NCCN) guidelines.
  Interventions: Combination Product: AZD4512 monotherapy
- Module 2 Dose Optimization (Experimental): Module 2 will randomize participants with R/R (as defined by NCCN guidelines) Ph(-) BALL only across 2 to 3 dose levels identified in Module 1 to receive AZD4512 monotherapy for further exploration of the doses. The aim of Module 2 is to identify the recommended Phase 2 dose (RP2D) of AZD4512 monotherapy, evaluate the efficacy and further define the safety profile of AZD4512.
  Interventions: Combination Product: AZD4512 monotherapy

INTERVENTIONS:
Combination Product: AZD4512 monotherapy — Patients will receive AZD4512 as monotherapy via intravenous infusion. AZD4512 is an antibody-drug conjugate targeting CD22

SUMMARY:
The study is intended to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of AZD4512 in patients with relapsed/refractory B-Cell acute lymphoblastic leukemia (r/r B-ALL).

DETAILED DESCRIPTION:
In this Phase I/II, open-label multi-center study AZD4512 will be administered to adult/young adult patients (Module 1: >=16 years; Module 2: >=12 years) with relapsed/refractory B-Cell acute lymphoblastic leukemia (B-ALL). This study will have 2 parts: Module 1 - Dose Escalation and Module 2 - Dose Optimization.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age:

  * 16 years old in Module 1
  * 12 years old in Module 2

    2. Diagnosis: Known Diagnosis of CD22-positive B-ALL based on criteria established by WHO (Alaggio et al. 2022).
* Participants must have relapsed or refractory B-ALL ('relapsed' defined as bone marrow blasts > 5% or reappearance of blasts in PB)
* Module 1 (DE): Ph(-) B-ALL and Ph(+) B-ALL - R/R
* Backfill of Module 1 and Module 2 (DO): R/R Ph(-) B-ALL (BM blasts >5%)

  3. Performance status (ECOG ≤ 2; KPS ≥ 50; LPS ≥ 50)

  4. Peripheral lymphoblast count < 10,000/µL (may receive cytoreduction prior to C1D1 per protocol-specified criteria)

  5. At least 2 prior therapies with refractoriness or relapse, or 1 prior therapy with refractoriness or relapse and no standard options available. Participants who have received prior CD22 targeted therapies are eligible.
* Ph+ B-ALL (Module 1 DE only): intolerant to or have contraindications to TKI therapy or R/R disease despite treatment with at least 2 prior TKIs or at least one 3rd generation TKI

  6. Prior DLI >4 weeks, prior cell therapy or autoHSCT >8 weeks, alloHSCT >12 weeks

Exclusion Criteria:

1. Burkitt lymphoma and leukemia
2. Isolated extramedullary disease; Active testicular or CNS (> CNS1) involvement
3. Unresolved non-heme toxicities Grade ≥ 2 (except alopecia, stable Grade ≤ 2 neuropathy, vitiligo, endocrine disorders controlled with therapy)
4. History of drug-induced non-infectious ILD/pneumonitis requiring oral or IV steroids or supplemental oxygen or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
5. Prior/concomitant therapy

   * Cytotoxic treatment within 14 days (except ALL maintenance medications or cytoreduction)
   * Biologic (immuno-oncology) treatment within 28 days or 5 half-lives (whichever is shorter)
   * Non-CNS radiation within 2 weeks & CNS radiation within 4 weeks
   * Medications known to prolong QTc and/or associated with Torsades de Pointes within 21 days or 5 half-lives (whichever is longer)
   * Strong inhibitors of CYP 3A4 within 21 days or 5 half-lives (whichever is longer)
   * Investigational agents or study interventions in the last 30 days or 5 half-lives prior to the first dose of AZD4512 whichever is longer. If the investigational product is an agent to treat B-ALL and meets the modality criteria, then a specific washout period must be adhered to instead.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Module 1 (Dose Escalation): Number of participants with dose-limiting toxicities (DLTs). | From first dose up to 21 days (DLT period).
  DLTs are dose-limiting toxicities as defined in the study protocol.
Module 1 (Dose Escalation): Frequency, duration and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  Assessed by the CTCAE criteria version 5.0
Module 1 (Dose Escalation): Frequency of dose interruptions, modifications, delays, and discontinuations due to AEs | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
Module 1 (Dose Escalation): Number of participants with clinically significant changes in laboratory values, ECGs, performance status, and vital signs | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
Module 2 (Dose Optimization): Overall response rate (ORR) in participants with R/R Ph(-) B-ALL | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy based on NCCN response criteria, measured by ORR (CR/CRh)
Module 2 (Dose Optimization): Frequency, duration and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  Assessed by the CTCAE criteria version 5.0
Module 2 (Dose Optimization): Frequency of dose interruptions, modifications, delays, and discontinuations due to AEs | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
Module 2 (Dose Optimization): Number of participants with clinically significant changes in laboratory values, ECGs, performance status, and vital signs | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)

SECONDARY OUTCOMES:
Module 1 (Dose Escalation): Plasma PK parameters of AZD4512 | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Total antibody and total unconjugated payload | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Area Under Curve (AUC) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Peak Plasma Concentration (Cmax) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Time to max concentration (Tmax) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Half life (T1/2) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Clearance (CL) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Volume of distribution (Vz) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Number and percentage of participants who develop anti-drug antibodies (ADAs) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To determine the immunogenicity of AZD4512 as monotherapy in participants with R/R B-ALL.
Module 1 (Dose Escalation): Objective Response Rate (ORR): proportion of participants with CR or CRh | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Composite Complete Remission (CRc) rate: proportion of participants with CR, CRh, or CRi | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Complete Remission (CR) rate | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Time to Response (TTR) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Duration of Response (DoR) | From date of first dose of AZD4512 up until end of study, up to 38 months
  - To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Event-Free Survival (EFS) | From date of first dose of AZD4512 up until end of study, up to 38 months
  - To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Overall Survival (OS) | From date of first dose of AZD4512 up until end of study, up to 38 months
  - To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 1 (Dose Escalation): Percentage of participants who receive subsequent allogeneic hematopoietic stem cell transplant (HSCT) | From date of first dose of AZD4512 up until end of study, up to 38 months
  - To evaluate the preliminary efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-) and Ph(+)] as defined by NCCN guidelines
Module 2 (Dose Optimization): Complete Remission (CR) rate | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization):Composite Complete Remission (CRc) rate: proportion of participants with CR, CRh, or CRi | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization):Time to Response (TTR) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization): Duration of Response (DoR) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization):Event-Free Survival (EFS) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization): Overall Survival (OS) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization): Percentage of participants who receive subsequent allogeneic hematopoietic stem cell transplant (HSCT) | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the efficacy of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)] as defined by NCCN guidelines
Module 2 (Dose Optimization): MRD-negative CR rate, CR/CRh (ORR), CR/CRi/CRh (CRc) rate | From date of first dose of AZD4512 up until end of study, up to 38 months
  To evaluate the impact of AZD4512 on MRD as assessed by NGS (central)
Module 2 (Dose Optimization): Plasma PK parameters of AZD4512 | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): total antibody and total unconjugated payload | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Area Under Curve (AUC) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimzation): Peak Plasma Concentration (Cmax) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Time to max concentration (Tmax) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Half life (T1/2) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Clearance (CL) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Volume of distribution (Vz) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To characterize the PK of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]
Module 2 (Dose Optimization): Summary of of pre-existing and treatment induced ADAs for AZD4512 (positive or negative, titers) | From date of first dose of AZD4512 up until 30 days post last dose of AZD4512 (on average 6 months)
  To determine the immunogenicity of AZD4512 as monotherapy in participants with R/R B-ALL [Ph(-)]

CONTACTS AND LOCATIONS:
Locations (23):
- United States (6):
  - Research Site, Duarte, California
  - Research Site, Jacksonville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Franklin, Tennessee
  - Research Site, Houston, Texas
- Research Site, Melbourne, Australia
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- China (2):
  - Research Site, Guangzhou
  - Research Site, Tianjin
- Japan (2):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, Bloomsbury
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/